## Midline Catheter Tip Positioning and Catheter-Related Complications during Antimicrobial Therapy: A Multicenter Randomized Controlled Trial

NCT04601597

**April 30, 2021** 

The current study followed the conformance study protocol analysis and conducted the statistical analysis using SAS 9.4 (http://www.sas.com/). The catheter measurement data were represented by mean and standard deviation according to the normal distribution. In contrast, the catheter measurement data with non-normal distribution were represented by median and quad, and the number of cases or percentages represented the counting data. The catheter-measurement data between the three groups were compared through variance analysis or the Kruskal-Wallis H test. Counting data were compared using the Chi-square test, exact probability method, and Kruskal-Wallis H test. The test level  $\alpha$ =0.05 for all three groups was a two-sided test, and P<0.05 was considered a statistically significant difference. Bonferroni method was used in pairwise comparison to optimize the significance level. The test levels α=0.017 and P<0.017 were statistically significant differences. To analyze the rate of complications, cumulative event rates were plotted as Kaplan-Meir curve, and differences in these rates were assessed using log-rank tests, and P<0.0001 was considered a statistically significant difference. Mann-Whitney U tests were performed to analyze the differences in observed event times.